CLINICAL TRIAL: NCT00858390
Title: Clinical Interventions to Increase Organ Procurement Nutritional Status and Enteral Absorption Capability After Brain Death (R38OT10585)
Brief Title: Nutritional Status and Enteral Absorption Capability After Brain Death
Acronym: HRSA Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Baylor College of Medicine (Other); LifeGift (Unknown)
Responsible Party: Principal Investigator, Georgene Hergenroeder, Assistant Professor, Neurosurgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R38OT10585; R38OT10585; HSC-MS-08-0473
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Brain Death
MeSH Terms: conditions — Brain Death | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 standard care (No Intervention): organ donors receiving standard care
- 2 Enteral Feeding (Experimental): enteral feeding with Oxepa® and RESOURCE® GLUTASOLVE®
  Interventions: Dietary Supplement: enteral feeding with Oxepa® and Glutasolve®

INTERVENTIONS:
Dietary Supplement: enteral feeding with Oxepa® and Glutasolve® — enteral feeding with Oxepa® and RESOURCE® GLUTASOLVE®
  Arms: 2 Enteral Feeding

SUMMARY:
The investigators propose to assess 36 donors' nutritional status using accepted parameters (prealbumin, resting energy expenditure); to assess nutrient intestinal absorption through 13Curacil breath tests; and to evaluate serum concentrations of IL-6 and TNFalpha to determine if continuing or initiating enteral feeding and nutritional supplementation is effective in restoring or maintaining nutritional parameters.

DETAILED DESCRIPTION:
There are an estimated 98,000 people in need of organ transplants in the United States (OPTN). Only a fraction of the need is met with the organs that become available. Therefore interventions are needed to maximize the viability of available organs and improve donor organ procurement and successful transplantation.

Improving the nutritional status of potential donors after they are declared brain dead could favorably impact subsequent organ procurement. Improved nutrition may improve organ viability by reducing the negative effects of inflammatory cytokines and catecholamines, and through reducing translocation of bacteria or endotoxin from the intestine.

In our preliminary work the investigators show significantly elevated inflammatory cytokines (IL-6 and TNFalpha) in unfed donors and a correlation with improved graft survival in recipients with lower plasma concentrations of IL-6.

The investigators propose to assess 36 donors' nutritional status using accepted parameters (prealbumin, resting energy expenditure); to assess nutrient intestinal absorption through 13Curacil breath tests; and to evaluate serum concentrations of IL-6 and TNFalpha to determine if continuing or initiating enteral feeding and nutritional supplementation is effective in restoring or maintaining nutritional parameters. Additionally, half of the group will be randomized to receive a nutritional supplement via naso/oro-duodenal feeding tube with a commercially available formula containing omega-3 and omega-6 fatty acids, and antioxidants plus glutamine (Oxepa® plus Glutasolve). The intervention through its anti-inflammatory and antioxidant functions has the potential to improve organ function (e.g. improved myocardial function (Wischmeyer 2003), and improved oxygenation (Pacht 2003; Pontes-Arruda 2006; Singer 2006)). Through improved organ function and/or a suppression of inflammatory cytokine production (e.g., IL-6 and TNFalpha) more organs are expected to be appropriate for procurement/transplantation.

If enteral nutrition reduces the inflammatory response commonly documented after brain death and, in doing so, improves organ procurement, enteral feeding could be immediately employed toward improving donor care practices. Furthermore, reducing the level of inflammatory molecules in donor organs may reduce the risk of rejection.

ELIGIBILITY:
Inclusion Criteria:

1. Consented solid organ donor
2. Age >14, <65 years old
3. Donors may have received or are receiving parenteral or enteral nutrition

Exclusion Criteria:

1. Known gastric or small bowel resections
2. Known malabsorptive disease of the gastrointestinal tract
3. Bariatric procedures, vagotomy or pyloroplasty
4. Known acute or chronic pancreatitis
5. Requiring an FiO2 > 60%

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-02; Primary Completion 2012-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgene Hergenroeder, MHA, RN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

REFERENCES:
- [Result] Hergenroeder GW, Ward NH, Yu X, Opekun A, Moore AN, Kozinetz CA, Powner DJ. Randomized trial to evaluate nutritional status and absorption of enteral feeding after brain death. Prog Transplant. 2013 Dec;23(4):374-82. doi: 10.7182/pit2013996. PMID 24311403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-six (36) brain dead organ donors were randomized in a 1:1 ratio to standard care (fasting) or to receive the nutritional intervention via naso/oro-duodenal feeding. Consent was obtained from family members for subject participation. Organ donors were screened and enrolled between 2/2009-6/2011.
Pre-assignment Details: Inclusion criteria: consented brain-dead organ donors age 14 to 70 years; may have received parenteral/enteral nutrition prior, but were excluded for prior gastric/bowel resections, GI malabsorption, bariatric procedures, vagotomy, pyloroplasty, or pancreatitis. Donors were excluded if a FiO2 greater than 60% was required (REE).
Groups:
- 1 Standard Care: 18 organ donors receiving standard care
- 2 Enteral Feeding: 18 enteral feeding with Oxepa® and RESOURCE® GLUTASOLVE®
  enteral feeding with Oxepa® and Glutasolve®: enteral feeding with Oxepa® and RESOURCE® GLUTASOLVE®
Period: Overall Study
Arm/Group | 1 Standard Care | 2 Enteral Feeding
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Standard Care | 2 Enteral Feeding | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (14.7) | 38.9 (14.5) | 41.9 (14.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 14 | 11 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 17 | 17 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 8 | 13 | 21
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36
Organs procured [Mean (Standard Deviation); unit: Solid organs procured] | 4.6 (1.5) | 4.4 (4.0) | 4.53 (1.7)
Organs Transplanted [Mean (Standard Deviation); unit: Solid organs transplanted] | 3.5 (1.8) | 4.1 (2.1) | 3.8 (2)
Positive Breath Test Results [Number; unit: participants] — An exhaled gas concentration of 9% cumulative percent dose recovery was defined as assimilating the 13C-uracil and therefore a positive breath test.
  participants | 4 | 6 | 10
Resting energy expenditure [Mean (Standard Deviation); unit: kcal/d] | 1954 (691.9) | 1773 (778.8) | 1866 (729.5)

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure is IL-6 Level
Description: Plasma IL-6 level measured by ELISA. The 12+/-2 hour time frame is prior to organ explantation.
Time Frame: 12+/-2 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | 1 Standard Care | 2 Enteral Feeding
Number analyzed (Participants) | 18 | 18
pg/ml | 565.5 (1010) | 264.9 (285.6)

ADVERSE EVENTS:
Arm/Group | 1 Standard Care | 2 Enteral Feeding
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This work was supported by the Department of Health and Human Services Health Resources and Services Administration Award Number 1R38OT10585-01-00 and, in part, by Public Health Service Grant DK56338.

Its contents are solely the responsibility of the authors and do not necessarily represent the official views of the PHS or HHS.